CLINICAL TRIAL: NCT04996004
Title: A Phase I/II Study of TTI-621 in Combination With Doxorubicin in Patients With Unresectable or Metastatic High-Grade Leiomyosarcoma
Brief Title: A Study to Learn About the Study Medicine (Called Ontorpacept or TTI-621) Given Alone and in Combination With Doxorubicin in People With Leiomyosarcoma
Acronym: TTI-621-03
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pfizer decided to terminate the study for administrative reasons. The termination was neither due to safety concerns nor a request from the regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTI-621-03; C4961003 (Other: Alias Study Number)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Leiomyosarcoma
Keywords: Leiomyosarcoma; Pleomorphic sarcoma; Myxofibrosarcoma; Liposarcoma; Angiosarcoma; Epithelioid sarcoma
MeSH Terms: conditions — Leiomyosarcoma; Dermatofibrosarcoma; Liposarcoma; Hemangiosarcoma; Sarcoma | interventions — TTI-621; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Ontorpacept+doxorubicin) (Experimental): In the dose escalation portion of the study, participants with specific subsets of soft tissue sarcomas who have not received more than one prior line of therapy and have not received an anthracycline in any setting will be enrolled in three escalating dose cohorts to characterize the safety and tolerability of Ontorpacept (TTI-621) when administered in combination with doxorubicin for up to six cycles and followed by Ontorpacept (TTI-621) monotherapy
  Interventions: Drug: Ontorpacept (TTI-621); Drug: Doxorubicin
- Dose Expansion Dose Level A (Cohort A) (Experimental): Participants with high-grade leiomyosarcoma will receive up to six cycles of Ontorpacept (TTI-621) at a pre-specified dose level (Dose Level A) in combination with fixed-dose doxorubicin followed by Ontorpacept (TTI-621) monotherapy to further characterize safety, tolerability, and clinical activity of the treatment regimen.
  Interventions: Drug: Ontorpacept (TTI-621); Drug: Doxorubicin
- Dose Expansion Dose Level B (Cohort B) (Experimental): Participants with high-grade leiomyosarcoma will receive up to six cycles of Ontorpacept (TTI-621) at a pre-specified dose level (Dose Level B) in combination with fixed-dose doxorubicin followed by Ontorpacept (TTI-621) monotherapy to further characterize safety, tolerability, and clinical activity of the treatment regimen.
  Interventions: Drug: Ontorpacept (TTI-621); Drug: Doxorubicin
- Dose Expansion Dose Level C (Cohort C) (Experimental): Participants with high-grade leiomyosarcoma will receive up to six cycles of Ontorpacept (TTI-621) at a pre-specified dose level (Dose Level C) in combination with fixed-dose doxorubicin followed by Ontorpacept (TTI-621) monotherapy to further characterize safety, tolerability, and clinical activity of the treatment regimen.
  Interventions: Drug: Ontorpacept (TTI-621); Drug: Doxorubicin

INTERVENTIONS:
Drug: Ontorpacept (TTI-621) — Ontorpacept (TTI-621) will be administered by intravenous infusion.
  Other Names: Ontorpacept / SIRPα-IgG1 Fc
Drug: Doxorubicin — 75 mg/m^2 by intravenous infusion in 21-day cycles for a maximum of six cycles.
  Other Names: Adriamycin

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (called Ontorpacept or TTI-621) when given alone and when given in combination with doxorubicin for people with leiomyosarcoma. Leiomyosarcoma is a tumor of the smooth muscles.

This study is seeking participants who have:

* leiomyosarcoma that is advanced or has spread to other parts of the body (metastatic)
* not received prior treatment with anthracyclines (a drug commonly used in patients with some kinds of cancer, including leiomyosarcoma)
* not received more than one prior treatment for their leiomyosarcoma During the first 18 weeks of this study, participants will receive doxorubicin by IV infusion (given directly into a vein) at the study clinic every 3 weeks for a total of 6 doses. Participants will also receive Ontorpacept (TTI-621) by IV infusion at the study clinic on the same day as doxorubicin and again one week later for the first 18 weeks.

After the first 18 weeks, participants will stop receiving doxorubicin but will continue receiving Ontorpacept (TTI-621) as IV infusion every 14 days at the study clinic. They will keep receiving Ontorpacept (TTI-621) until their cancer is no longer responding to treatment.

We will examine the experiences of participants receiving Ontorpacept (TTI-621) in combination with doxorubicin in the first 18 weeks and then Ontorpacept (TTI-621) by itself after the doxorubicin is stopped. This will help us determine if the study medicine Ontorpacept (TTI-621) given with doxorubicin and then by itself is safe and effective.

Participants will be involved in the study for approximately one year, depending on how their cancer responds to the study treatment. They will have study visits about 12 times in the first 18 weeks (when the study medicine Ontorpacept is given with doxorubicin) and then every two weeks after the doxorubicin is stopped and the study medicine Ontorpacept (TTI-621) is given by itself.

DETAILED DESCRIPTION:
This trial will be conducted in 2 phases: Phase I (dose escalation of Ontorpacept in combination with fixed-dose doxorubicin) and Phase II (dose expansion of Ontorpacept in combination with fixed-dose doxorubicin).

Phase I will enroll patients with soft-tissue sarcomas including leiomyosarcoma, undifferentiated pleomorphic sarcoma, myxofibrosarcoma, dedifferentiated liposarcoma, angiosarcoma or epithelioid sarcoma to evaluate escalating doses of Ontorpacept (TTI-621) administered in combination with fixed-dose doxorubicin for up to six cycles followed by Ontorpacept (TTI-621) monotherapy.

Phase II will enroll patients with high-grade leiomyosarcoma and will evaluate two dose levels of Ontorpacept (TTI-621) in combination with fixed-dose doxorubicin for up to six cycles followed by Ontorpacept (TTI-621) monotherapy.

.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Co-operative Oncology Group Performance Status Performance Status (ECOG-PS) 0 or 1.
2. Histologically-confirmed high-grade soft tissue sarcoma that is metastatic or locally advanced and not amenable to curative treatment with surgery or radiation.

   1. In the Dose Escalation phase, indications will be limited to high-grade leiomyosarcoma, undifferentiated pleomorphic sarcoma, myxofibrosarcoma, dedifferentiated liposarcoma, angiosarcoma and epithelioid sarcoma
   2. In the Dose Expansion phase, indications will be limited to high-grade leiomyosarcoma.
3. Objective evidence of disease progression unless disease is newly-diagnosed.
4. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (expansion cohorts).
5. Adequate organ and hematologic function.
6. No more than 1 prior treatment regimen for advanced disease, which is limited to gemcitabine with docetaxel.
7. Anthracycline-naïve.
8. Patients who were treated with a prior chemotherapy regimen must have completed treatment at least three weeks before initiation of study treatment.
9. All adverse events from prior treatment must be NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v5 Grade ≤ 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline.
10. Radiotherapy, including palliative radiotherapy, completed at least two weeks prior to treatment; palliative radiation to non-target lesions while on study is allowed.

Key Exclusion Criteria:

1. History of acute coronary syndromes.
2. History of or current Class II, III, or IV heart failure.
3. History or evidence of known CNS (central nervous system) metastases or carcinomatous meningitis.
4. Significant bleeding disorders, vasculitis or a significant bleeding episode from the GI (gastrointestinal) tract.
5. History of severe hypersensitivity reactions to antibodies.
6. Systemic steroid therapy.
7. History or autoimmune disease that has required systemic treatment with disease-modifying agents, corticosteroids, or immunosuppressive drugs.
8. Prior organ transplantation including allogenic or autologous stem cell transplantation
9. Prior treatment with anti-CD47 (Cluster of Differentiation 47) or anti-signal regulatory protein alpha (SIRPα) therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - MSK Basking Ridge., Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack., Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center 53rd street., New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - MSK Nassau, Uniondale, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Oregon Health and Science University - Center for Health and Healing 1 (CHH1), Portland, Oregon
  - Oregon Health and Science University - Center for Health and Healing 2(CHH2), Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TTI-621-03

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of two phases: Phase I (dose escalation) and Phase II (dose expansion). Phase I enrolled participants with high-grade leiomyosarcoma, undifferentiated pleomorphic sarcoma, myxofibrosarcoma, dedifferentiated liposarcoma, angiosarcoma and epithelioid sarcoma. Phase II enrolled participants with high-grade leiomyosarcoma. Participants were treated with ontorpacept (TTI-621) in combination with doxorubicin for the first 6 cycles and ontorpacept alone thereafter.
Pre-assignment Details: A total of 76 participants were enrolled and treated in the study (Phase I: 9 participants and Phase II: 67 participants).
Groups:
- Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin: Participants received ontorpacept, 0.2 milligram per kilogram (mg/kg) as Intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 milligram per meter square (mg/m^2) was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 0.2 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
- Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin: Participants received ontorpacept, 0.7 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 0.7 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
- Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin; Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B): Participants received ontorpacept, 2.0 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 2.0 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
- Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A): Participants received ontorpacept, 0.2 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 0.2 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
- Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C): Participants received ontorpacept, 1.0 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 1.0 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
Period: Phase I
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Started | 3 | 3 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 2 | 1 | 2 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Started | 0 | 0 | 0 | 32 | 13 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 32 | 13 | 22
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 20 | 10 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 12 | 2 | 9
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment.
Groups:
- Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin; Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A): Participants received ontorpacept, 0.2 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 0.2 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
- Total: Total of all reporting groups
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22 | 76
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 40 years | 1 | 0 | 0 | 3 | 1 | 0 | 5
  40 - <65 years | 2 | 1 | 2 | 25 | 7 | 12 | 49
  65 - <75 years | 0 | 1 | 1 | 4 | 5 | 7 | 18
  75 - <85 years | 0 | 1 | 0 | 0 | 0 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 23 | 10 | 16 | 55
  Male | 1 | 2 | 0 | 9 | 3 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 2 | 2 | 2 | 9
  Not Hispanic or Latino | 2 | 2 | 2 | 29 | 10 | 19 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 0 | 0 | 3
  White | 2 | 3 | 3 | 24 | 10 | 22 | 64
  More than one race | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs: Phase I
Description: An adverse event (AE) was any untoward medical occurrence or worsening of a pre-existing medical condition following or during exposure to pharmaceutical product, whether or not considered causally related to product. A serious adverse event (SAE) was an adverse event occurred during any study at any dose of the investigational products that fulfils one or more of following criteria: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. TEAEs were those events with onset date occurred during on-treatment period. AEs included SAEs and all Non-SAEs. On-treatment period was defined as time from first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer therapy). Participant with at least one TEAE and one serious TEAEs are reported in this outcome measure.
Time Frame: From first dose of study treatment (Day 1) up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure for Phase I was 74.1 weeks; maximum follow up to approx. 78.1 weeks)
Population: The safety analysis set (SAS) included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Participants with TEAEs | 3 | 3 | 3
  Participants with Serious TEAEs | 0 | 1 | 1

2. Primary Outcome: Mean Change From Baseline in Blood Pressure at 30 Minutes Post Dose on Cycle 1 Day 1 (C1D1): Phase I
Description: Blood pressure included diastolic blood pressure (DBP) and systolic blood pressure (SBP). Mean change from baseline to 30 minutes post-dose on C1D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 30 minutes post dose on Day 1 of Cycle 1
Population: The SAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Millimeter of mercury (mmHg)
  DBP | -0.7 (5.86) | -0.7 (3.51) | 1.0 (8.72)
  SBP | 1.7 (8.02) | 2.0 (3.61) | -8.7 (4.73)

3. Primary Outcome: Mean Change From Baseline in Blood Pressure at 60 Minutes Post Dose on C1D1: Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 60 minutes post-dose on C1D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 60 minutes post dose on Day 1 of Cycle 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Millimeter of mercury
  DBP | 2.3 (2.08) | 0.7 (3.21) | 1.7 (9.29)
  SBP | 3.0 (5.00) | -0.7 (2.89) | -8.3 (10.12)

4. Primary Outcome: Mean Change From Baseline in Blood Pressure at 30 Minutes Post Dose on Cycle 1 Day 8 (C1D8): Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 30 minutes post-dose on C1D8 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 30 minutes post dose on Day 8 of Cycle 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Millimeter of mercury
  DBP | 1.3 (10.02) | 2.7 (5.03) | 0.3 (2.89)
  SBP | 7.0 (11.36) | 5.0 (6.93) | -7.3 (7.51)

5. Primary Outcome: Mean Change From Baseline in Blood Pressure at 60 Minutes Post Dose on C1D8: Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 60 minutes post-dose on C1D8 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 60 minutes post dose on Day 8 of Cycle 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Groups:
- Phase I : Ontorpacept 0.7 mg/kg + Doxorubicin: Participants received ontorpacept, 0.7 mg/kg as IV infusion on Days 1 and 8 of each 21-day cycle up to Cycle 6. Doxorubicin 75 mg/m^2 was administered as IV infusion on Day 1 of 21-day cycles for a maximum of 6 cycles. After Cycle 6, participants continued treatment with ontorpacept 0.7 mg/kg as IV infusion on Days 1 and 15 as monotherapy in 28-day cycles until documentation of disease progression or development of unacceptable toxicity and a long-term follow-up period for assessment of overall survival.
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I : Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Millimeter of mercury
  DBP | 0.3 (9.81) | -4.0 (7.94) | 0.7 (6.51)
  SBP | 3.3 (9.07) | 2.3 (9.29) | -1.0 (11.53)

6. Primary Outcome: Mean Change From Baseline in Blood Pressure at 30 Minutes Post Dose on Cycle 2 Day 1 (C2D1): Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 30 minutes post-dose on C2D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 30 minutes post dose on Day 1 of Cycle 2
Population: The SAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 2
Millimeter of mercury
  DBP | 3.0 (3.46) | -2.0 (6.24) | 6.5 (3.54)
  SBP | 4.0 (5.29) | -5.7 (6.51) | 3.5 (16.26)

7. Primary Outcome: Mean Change From Baseline in Blood Pressure at 60 Minutes Post Dose on C2D1: Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 60 minutes post-dose on C2D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 60 minutes post dose on Day 1 of Cycle 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 2
Millimeter of mercury
  DBP | 3.0 (5.20) | -3.7 (8.02) | 11.0 (1.41)
  SBP | 5.0 (5.57) | -2.0 (14.73) | 10.5 (24.75)

8. Primary Outcome: Mean Change From Baseline in Blood Pressure at 30 Minutes Post Dose on Cycle 3 Day 1 (C3D1): Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 30 minutes post-dose on C3D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 30 minutes post dose on Day 1 of Cycle 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 2 | 1
Millimeter of mercury
  DBP | -3.5 (6.36) | -5.5 (4.95) | 2.0 (NA) — Standard deviation (SD) could not be calculated as only 1 participant was analyzed.
  SBP | -6.5 (17.68) | -14.0 (0.00) | -8.0 (NA) — SD could not be calculated as only 1 participant was analyzed.

9. Primary Outcome: Mean Change From Baseline in Blood Pressure at 60 Minutes Post Dose on C3D1: Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to 60 minutes post-dose on C3D1 were reported in this outcome measure. Baseline was defined as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, 60 minutes post dose on Day 1 of Cycle 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 2 | 1
Millimeter of mercury
  DBP | 0.5 (6.36) | -2.0 (2.83) | 6.0 (NA) — SD could not be calculated as only 1 participant was analyzed.
  SBP | -1.0 (7.07) | -12.0 (4.24) | -11.0 (NA) — SD could not be calculated as only 1 participant was analyzed.

10. Primary Outcome: Mean Change From Baseline in Blood Pressure at Safety Follow up: Phase I
Description: Blood pressure included DBP and SBP. Mean change from baseline to safety follow up visit were reported in this outcome measure. Baseline was considered as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, Safety follow up (up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure for Phase I was 74.1 weeks; maximum follow up to approx. 78.1 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 3 | 3
Millimeter of mercury
  DBP | 7.0 (2.83) | -10.3 (2.89) | 3.0 (13.08)
  SBP | 13.5 (14.85) | -15.7 (10.07) | 8.7 (12.66)

11. Primary Outcome: Mean Change From Baseline in Body Weight at C3D1: Phase I
Description: Body weight was measured in kilograms (kg). Baseline was considered as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, Day 1 of Cycle 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 2 | 2
Kilograms | 0.68 (0.962) | -3.86 (2.885) | -1.71 (0.148)

12. Primary Outcome: Mean Change From Baseline in Body Weight at Cycle 5 Day 1 (C5D1): Phase I
Description: Body weight was measured in kilograms. Baseline was considered as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1).
Time Frame: Baseline, Day 1 of Cycle 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 2 | 2
Kilograms | -0.91 (0.000) | -2.50 (5.452) | -2.09 (1.534)

13. Primary Outcome: Mean Change From Baseline in Body Weight at Cycle 7 Day 1 (C7D1): Phase I
Description: as for outcome 12
Time Frame: Baseline, Day 1 of Cycle 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 2 | 2
Kilograms | -0.91 (0.636) | -0.23 (2.249) | -1.26 (0.785)

14. Primary Outcome: Mean Change From Baseline in Body Weight at Safety Follow up: Phase I
Description: as for outcome 12
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 2 | 3 | 3
kilograms | 1.13 (0.325) | -3.48 (1.889) | -1.56 (1.794)

15. Primary Outcome: Number of Participants With Overall Electrocardiogram (ECG) Abnormalities: Phase I
Description: Standard 12- lead ECGs, average of triplicate assessments were obtained in participant in supine position and within 10 minutes total time. ECG abnormalities included: PR interval (millisecond [msec]): value greater than or equal to (>=) 220 and change from baseline >=20; QRS interval (msec) value >=120; uncorrected QT interval, QT correct by Bazzette's formula (QTcB) interval and QT correct by Frederica formula (QTcF) interval (msec): value greater than (>) 450, value > 480, value > 500, change from baseline > 30 and > 60. Baseline was defined as the last assessment prior to the date or time of the first dose of study treatment. In this outcome measure number of participants with overall ECG abnormalities are reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants | 3 | 2 | 2

16. Primary Outcome: Number of Participants With Shift in National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v)5.0 Grade <=2 at Baseline to >=3 Post-baseline in Hematology Parameters: Phase I
Description: The following hematology laboratory parameters were assessed: hemoglobin, hematocrit, platelets, white blood cells (WBC), neutrophils, lymphocytes, eosinophils, basophils, monocytes, WBC with automated 5-part differential, Red blood cells (RBC), absolute reticulocytes, reticulocytes percentage (%), Mean corpuscular hemoglobin (MCH), Mean corpuscular volume (MCV) and Red cell distribution width (RDW). Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. Baseline was defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants who had hematology parameter abnormality Grade <=2 at baseline and shifted to >=3 post-baseline are reported in this outcome measure. Only non-zero categories for any reporting arm are reported.
Time Frame: Baseline up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure for Phase I was 74.1 weeks; maximum follow up to approx. 78.1 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Shift from baseline Grade to post-baseline Grade 3: Leukocytes (10^9/L) white blood cells decreased | 1 | 2 | 1
  Shift from baseline Grade to post-baseline Grade 4: Leukocytes (10^9/L) white blood cells decreased | 0 | 0 | 2
  Shift from baseline Grade to post-baseline Grade 3: Neutrophils (10^9/L) decreased | 1 | 1 | 0
  Shift from baseline Grade to post-baseline Grade 4: Neutrophils (10^9/L) decreased | 0 | 0 | 3
  Shift from baseline Grade to post-baseline Grade 3: Platelets (10^9/L) decreased | 0 | 1 | 2

17. Primary Outcome: Number of Participants With Shift in NCI-CTCAE v5.0 Grade <=2 at Baseline to >=3 Post-baseline in Chemistry Parameters: Phase I
Description: The following chemistry parameters were assessed: glucose, sodium, potassium, calcium, chloride, phosphate, bicarbonate, blood urea nitrogen or urea, creatinine, total protein, albumin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, indirect bilirubin, uric acid, calcium, magnesium, lactate dehydrogenase (LDH). Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death related to adverse event. Baseline was defined as last assessment prior to date/time of first dose of study treatment. Number of participants who had chemistry parameter abnormality Grade<=2 at baseline and shifted to >=3 post-baseline are reported in this outcome measure. Only non-zero categories for any reporting arm are reported.
Time Frame: as for outcome 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Shift from baseline Grade to post-baseline Grade 3: ALT (U/L) increased | 0 | 1 | 0
  Shift from baseline Grade to post-baseline Grade 4: AST (U/L) increased | 0 | 1 | 0

18. Primary Outcome: Number of Participants With Dose Modifications: Phase I
Description: Dose modifications included dose reduction, dose omitted, infusion interruption and cycle delayed.
Time Frame: During study treatment (from first dose of study treatment [Day 1] to maximum treatment exposure of 74.1 weeks for ontorpacept and 20.1 weeks for doxorubicin)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Participants with dose reduction- Ontorpacept | 0 | 0 | 0
  Participants with dose omitted- Ontorpacept | 0 | 1 | 2
  Participants with infusion interruption-Ontorpacept | 0 | 1 | 1
  Participants with cycle delayed- Ontorpacept | 1 | 1 | 0
  Participants with dose reduction- Doxorubicin | 0 | 1 | 2
  Participants with dose omitted- Doxorubicin | 0 | 0 | 0
  Participants with infusion interruption-Doxorubicin | 0 | 0 | 0
  Participants with cycle delayed- Doxorubicin | 1 | 0 | 0

19. Primary Outcome: Number of Participants With Treatment Discontinuations: Phase I
Description: Number of participants with treatment discontinuations during the study treatment were reported in this outcome measure.
Time Frame: as for outcome 18
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Ontorpacept | 3 | 3 | 3
  Doxorubicin | 1 | 2 | 2

20. Primary Outcome: Objective Response Rate (ORR): Phase I and Phase II
Description: ORR: percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on investigator's assessment per response evaluation criteria in solid tumours RECIST version (v)1.1. BOR: best response recorded from start of treatment until disease progression (PD). CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than(< )10 mm. PR: at least 30 percent (%) decrease in sum of longest diameter of target lesions, taking as reference baseline sum longest diameter. PD: at least 20% increase in sum of longest diameter of target lesions, taking as reference of the smallest sum on study.
Time Frame: From the start of study treatment until disease progression (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: The FAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Percentage of Participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 18.8 [7.2 to 36.4] | 0.0 [0.0 to 24.7] | 4.5 [0.1 to 22.8]

21. Secondary Outcome: Number of Participants With TEAEs and Serious TEAEs: Phase II
Description: An AE was any untoward medical occurrence or worsening of a pre-existing medical condition following or during exposure to pharmaceutical product, whether or not considered causally related to product. A SAE was an adverse event occurred during any study at any dose of the investigational products that fulfils one or more of following criteria: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. TEAEs were those events with onset date occurred during on-treatment period. AEs included SAEs and all Non-SAEs. On-treatment period was defined as time from first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer therapy). Participant with at least one TEAE and one serious TEAEs are reported in this outcome measure.
Time Frame: From first dose of study treatment (Day 1) up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure for Phase II was 88 weeks; maximum follow up to approx. 92 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants
  Participants with TEAEs | 32 | 13 | 22
  Participants with Serious TEAEs | 9 | 8 | 15

22. Secondary Outcome: Mean Change From Baseline in Blood Pressure: Phase II
Description: as for outcome 10
Time Frame: Baseline, 30 and 60min post dose of C1D1,C1D8,C2D1,C3D1 and safety follow up 30 Days post last dose of study treatment/start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure of Phase II:88 weeks;maximum follow up:92 weeks)
Population: The SAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Millimeter of mercury
  DBP: Change at 30 minutes post dose on C1D1: number analyzed (Participants) | 27 | 13 | 20
  DBP: Change at 30 minutes post dose on C1D1 | -2.8 (7.46) | -8.8 (5.37) | -3.5 (11.31)
  DBP: Change at 60 minutes post dose on C1D1: number analyzed (Participants) | 24 | 13 | 19
  DBP: Change at 60 minutes post dose on C1D1 | -1.4 (6.73) | -7.8 (7.01) | -4.5 (11.88)
  SBP: Change at 30 minutes post dose on C1D1: number analyzed (Participants) | 27 | 13 | 20
  SBP: Change at 30 minutes post dose on C1D1 | -10.0 (12.82) | -15.4 (15.06) | -3.6 (14.04)
  SBP: Change at 60 minutes post dose on C1D1: number analyzed (Participants) | 24 | 13 | 19
  SBP: Change at 60 minutes post dose on C1D1 | -5.0 (12.18) | -18.3 (15.70) | -6.5 (14.79)
  DBP: Change at 30 minutes post dose on C1D8: number analyzed (Participants) | 21 | 6 | 4
  DBP: Change at 30 minutes post dose on C1D8 | -3.5 (10.78) | -5.0 (6.63) | 6.3 (15.26)
  DBP: Change at 60 minutes post dose on C1D8: number analyzed (Participants) | 20 | 6 | 3
  DBP: Change at 60 minutes post dose on C1D8 | -1.8 (9.08) | -4.8 (5.81) | 1.7 (2.52)
  SBP: Change at 30 minutes post dose on C1D8: number analyzed (Participants) | 21 | 6 | 4
  SBP: Change at 30 minutes post dose on C1D8 | -9.0 (14.23) | -7.0 (16.52) | 15.5 (20.14)
  SBP: Change at 60 minutes post dose on C1D8: number analyzed (Participants) | 20 | 6 | 3
  SBP: Change at 60 minutes post dose on C1D8 | -6.8 (12.26) | -9.5 (14.54) | 11.7 (8.96)
  DBP: Change at 30 minutes post dose on C2D1: number analyzed (Participants) | 13 | 4 | 9
  DBP: Change at 30 minutes post dose on C2D1 | -3.3 (6.58) | 0.8 (8.30) | -7.6 (15.95)
  DBP: Change at 60 minutes post dose on C2D1: number analyzed (Participants) | 12 | 4 | 8
  DBP: Change at 60 minutes post dose on C2D1 | -3.8 (7.27) | -3.5 (8.23) | -3.1 (13.36)
  SBP: Change at 30 minutes post dose on C2D1: number analyzed (Participants) | 13 | 4 | 9
  SBP: Change at 30 minutes post dose on C2D1 | -9.1 (14.57) | -3.3 (19.29) | -9.9 (17.51)
  SBP: Change at 60 minutes post dose on C2D1: number analyzed (Participants) | 12 | 4 | 8
  SBP: Change at 60 minutes post dose on C2D1 | -7.7 (11.62) | -11.5 (5.80) | -6.3 (13.41)
  DBP: Change at 30 minutes post dose on C3D1: number analyzed (Participants) | 10 | 4 | 4
  DBP: Change at 30 minutes post dose on C3D1 | -4.4 (4.09) | -6.8 (13.02) | -2.3 (6.50)
  DBP: Change at 60 minutes post dose on C3D1: number analyzed (Participants) | 10 | 4 | 3
  DBP: Change at 60 minutes post dose on C3D1 | -3.2 (6.16) | -10.0 (9.90) | -2.0 (1.00)
  SBP: Change at 30 minutes post dose on C3D1: number analyzed (Participants) | 10 | 4 | 4
  SBP: Change at 30 minutes post dose on C3D1 | -14.1 (12.20) | -7.3 (10.66) | -7.3 (20.50)
  SBP: Change at 60 minutes post dose on C3D1: number analyzed (Participants) | 10 | 4 | 3
  SBP: Change at 60 minutes post dose on C3D1 | -14.3 (13.37) | -11.8 (5.74) | -8.0 (17.44)
  DBP: Change at safety follow up: number analyzed (Participants) | 27 | 7 | 15
  DBP: Change at safety follow up | -2.3 (12.10) | -1.3 (13.52) | 2.1 (12.95)
  SBP: Change at safety follow up: number analyzed (Participants) | 27 | 7 | 15
  SBP: Change at safety follow up | -6.9 (16.86) | -2.4 (26.30) | 0.2 (16.11)

23. Secondary Outcome: Mean Change From Baseline in Body Weight: Phase II
Description: Baseline was considered as the last measurement taken prior to the first infusion of study medication (Day 1 of Cycle 1)
Time Frame: Baseline, Day 1 of Cycle 3, 5, 7 and safety follow up (up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest [maximum treatment exposure for Phase II was 88 weeks; maximum follow up to 92 weeks])
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Kilograms
  Change at C3D1: number analyzed (Participants) | 25 | 11 | 14
  Change at C3D1 | -1.30 (1.765) | -0.43 (2.122) | -1.83 (1.637)
  Change at C5D1: number analyzed (Participants) | 23 | 8 | 14
  Change at C5D1 | -1.23 (2.348) | -1.03 (2.807) | -2.44 (2.620)
  Change at C7D1: number analyzed (Participants) | 22 | 5 | 11
  Change at C7D1 | -0.84 (2.836) | 1.03 (2.420) | -2.57 (3.695)
  Change at Follow up: number analyzed (Participants) | 27 | 6 | 13
  Change at Follow up | -0.54 (3.757) | 0.18 (3.012) | -3.55 (5.018)

24. Secondary Outcome: Number of Participants With Overall ECG Abnormalities: Phase II
Description: Standard 12- lead ECGs, average of triplicate assessments was obtained in participant in supine position and within 10 minutes total time. ECG abnormalities included: PR interval (msec): >= 220 and change from baseline >=20; QRS interval (msec) value >=120; uncorrected QT interval, QT correct by QTcB interval and QT correct by QTcF interval (msec): value > 450, value > 480, value > 500, change from baseline > 30 and > 60. Baseline was defined as the last assessment prior to the date or time of the first dose of study treatment. In this outcome measure number of participants with overall ECG abnormalities are reported.
Time Frame: as for outcome 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants | 17 | 8 | 11

25. Secondary Outcome: Number of Participants With Shift in NCI-CTCAE v5.0 Grade <=2 at Baseline to >=3 Post-baseline in Hematology Parameters: Phase II
Description: The following hematology laboratory parameters were assessed: hemoglobin, hematocrit, platelets, WBC, neutrophils, lymphocytes, eosinophils, basophils, monocytes, WBC with automated 5-part differential, RBC, absolute reticulocytes, reticulocytes %, MCH, MCV and RDW. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. Baseline was defined as the last assessment prior to the date/time of the first dose of study treatment. Number of participants who had hematology parameter abnormality Grade <=2 at baseline and shifted to >=3 post-baseline are reported in this outcome measure. Only non-zero categories for any reporting arm are reported.
Time Frame: Baseline up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurred soonest (maximum treatment exposure for Phase II was 88 weeks; maximum follow up to approx. 92 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants
  Shift from baseline Grade to post-baseline Grade 3: Leukocytes (10^9/L) white blood cells decreased | 12 | 3 | 7
  Shift from baseline Grade to post-baseline Grade 4: Leukocytes (10^9/L) white blood cells decreased | 12 | 9 | 12
  Shift from baseline Grade to post-baseline Grade 3: Neutrophils (10^9/L) decreased | 5 | 2 | 6
  Shift from baseline Grade to post-baseline Grade 4: Neutrophils (10^9/L) decreased | 21 | 10 | 8
  Shift from baseline Grade to post-baseline Grade 3: Platelets (10^9/L) decreased | 4 | 6 | 12
  Shift from baseline Grade to post-baseline Grade 4: Platelets (10^9/L) decreased | 2 | 1 | 7

26. Secondary Outcome: Number of Participants With Shift in NCI-CTCAE v5.0 Grade <=2 at Baseline to >=3 Post-baseline in Chemistry Parameters: Phase II
Description: The following chemistry parameters were assessed: glucose, sodium, potassium, calcium, chloride, phosphate, bicarbonate, blood urea nitrogen or urea, creatinine, total protein, albumin, alkaline phosphatase, AST, ALT, total bilirubin, indirect bilirubin, uric acid, calcium, magnesium and LDH. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death related to adverse event. Baseline was defined as last assessment prior to date/time of first dose of study treatment. Number of participants who had chemistry parameter abnormality Grade<=2 at baseline and shifted to >=3 post-baseline are reported in this outcome measure. Only non-zero categories for any reporting arm are reported.
Time Frame: as for outcome 25
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants
  Shift from baseline Grade to post-baseline Grade 3: ALT (U/L) increased | 0 | 0 | 1
  Shift from baseline Grade to post-baseline Grade 3: Albumin; Hypoalbuminemia (g/L) | 0 | 0 | 1
  Shift from baseline Grade to post-baseline Grade 3: Blood Bilirubin increased (umol/L) | 0 | 1 | 0
  Shift from baseline Grade to post-baseline Grade 3: Magnesium; Hypermagnesemia (mmol/L) | 1 | 0 | 1

27. Secondary Outcome: Number of Participants With Dose Modifications: Phase II
Description: Dose modifications included dose reduction, dose omitted, infusion interruption and cycle delayed.
Time Frame: During study treatment (from first dose of study treatment [Day 1] to maximum treatment exposure of 88 weeks for ontorpacept and 25 weeks for doxorubicin)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants
  Participants with dose reduction- Ontorpacept | 0 | 5 | 17
  Participants with dose omitted- Ontorpacept | 14 | 7 | 19
  Participants with infusion interruption- Ontorpacept | 2 | 7 | 11
  Participants with cycle delayed- Ontorpacept | 15 | 5 | 5
  Participants with dose reduction- Doxorubicin | 11 | 5 | 13
  Participants with dose omitted- Doxorubicin | 1 | 0 | 3
  Participants with infusion interruption- Doxorubicin | 0 | 1 | 0
  Participants with cycle delayed- Doxorubicin | 8 | 4 | 2

28. Secondary Outcome: Number of Participants With Treatment Discontinuations: Phase II
Description: Number of participants with treatment discontinuations during the study treatment were reported in this outcome measure.
Time Frame: as for outcome 27
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 32 | 13 | 22
Participants
  Ontorpacept | 32 | 13 | 22
  Doxorubicin | 15 | 5 | 10

29. Secondary Outcome: Progression Free Survival (PFS): Phase I and Phase II
Description: PFS was defined as the time from the first ontorpacept infusion (Day 1 of Cycle 1) to PD or death of any cause, whichever occurred first. PD was defined at least 20% increase in sum of longest diameter (LD) of target lesion, taking reference of smallest sum on study. Participants without PD or death or participants with an event after 2 or more missing/inadequate disease assessment or participants with an event after the start date of alternate anticancer therapy were censored at their last response assessment date or last assessment prior to the start date of alternate anti-cancer therapy, whichever is earlier. Kaplan-Meier method was used for analysis.
Time Frame: Time from the first ontorpacept infusion (Day 1 of Cycle 1) to PD or death of any cause or censoring, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Months | 7.9 [1.2 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated due to insufficient number of participants with events. | 6.4 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.6 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 6.0 [4.1 to 6.7] | 4.3 [1.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 5.6 [3.0 to 9.7]

30. Secondary Outcome: Overall Survival (OS): Phase I and Phase II
Description: OS was defined as the time from the first ontorpacept infusion (Day 1 of Cycle 1) to death of any cause. Participants last known to be alive were censored at their last known alive date. Kaplan-Meier method was used for analysis.
Time Frame: From the first ontorpacept infusion (Day 1 of Cycle 1) to death of any cause or censoring, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Months | NA [26.0 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 8.2 [7.2 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [4.1 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 20.5 [15.7 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [4.9 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 14.4 [12.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

31. Secondary Outcome: Disease Control Rate (DCR): Phase I and Phase II
Description: DCR was defined as the percentage of participants who have achieved CR, PR, or SD lasting at least 4 weeks as per RECIST v1.1 CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: at least 30% decrease in sum of longest diameter of target lesions, taking as reference baseline sum longest diameter. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum LD since treatment started. PD: at least 20% increase in sum of longest diameter of target lesions, taking as reference of the smallest sum on study.
Time Frame: From the first dose of study treatment until PD or death, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Percentage of participants | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 75.0 [56.6 to 88.5] | 84.6 [54.6 to 98.1] | 72.7 [49.8 to 89.3]

32. Secondary Outcome: Duration of Response (DOR): Phase I and Phase II
Description: DOR was defined as time from date of first documented response (CR or PR) to date of documented progression or death of any cause after achieving response. DOR was calculated for participants who achieved CR or PR. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: at least 30% decrease in sum of longest diameter of target lesions, taking as reference baseline sum longest diameter. Participants without PD or death or participants with an event after 2 or more missing/inadequate disease assessment or participants with an event after the start date of alternate anticancer therapy were censored at their last response assessment date or last assessment prior to the start date of alternate anti-cancer therapy, whichever is earlier.
Time Frame: Time from date of first documented response (CR or PR) to date of documented progression or death of any cause after achieving response or censoring, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: The FAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment. Here "Number of Participants Analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 0 | 0 | 1 | 6 | 0 | 1
Months |  |  | 9.7 [NA to NA] — Full range of 95% CI could not be calculated as only one participant was evaluable. | 4.7 [3.5 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. |  | NA [NA to NA] — Median and full range of 95% CI could not be calculated as participant did not have event of interest.

33. Secondary Outcome: Duration of Disease Control (DDC): Phase I and Phase II
Description: DDC: participants who achieved BOR of SD, as time from first ontorpacept infusion (Day1 of Cycle1) to date of documented PD/death of any cause. Calculated for participants who achieved CR,PR/SD lasting at least 4weeks. CR:disappearance of all target lesion. Any pathological lymph nodes must have reduction in short axis to<10 mm. PR:at least 30%decrease in sum of longest diameter of target lesions, taking as reference baseline sum longest diameter. SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum LD since treatment started. PD:at least 20% increase in sum of LD of target lesion, taking reference of smallest sum on study. Participants without PD/death/with an event after 2/more missing/inadequate disease assessment/with event after start date of alternate anticancer therapy were censored at last response assessment date/last assessment prior to start date of alternate anti-cancer therapy, whichever is earlier.
Time Frame: Time from first ontorpacept infusion (Day 1 of Cycle 1) to date of documented progression/death of any cause or censoring, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: The FAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 2 | 2 | 2 | 24 | 11 | 16
Months | 12.4 [7.9 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [6.4 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 10.6 [7.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 6.1 [5.9 to 9.7] | 4.7 [2.1 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 6.1 [4.1 to 11.8]

34. Secondary Outcome: Time to Progression (TTP): Phase I and Phase II
Description: TTP was defined as the time from the first ontorpacept infusion (Day 1 of Cycle 1) to PD or death of any cause, whichever is first; provided death was not considered as an event. PD: at least 20% increase in sum of longest diameter of target lesion, taking reference of smallest sum on study. Participants without PD or death or with an event after 2 or more missing or inadequate disease assessment or with event after start date of alternate anticancer therapy were censored at last response assessment date or last assessment prior to start date of alternate anti-cancer therapy, whichever is earlier.
Time Frame: Time from the first ontorpacept infusion (Day 1 of Cycle 1) to PD or death of any cause or censoring, whichever is first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Months | 7.9 [1.2 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 6.4 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.6 [1.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 6.0 [4.2 to 6.7] | 4.3 [1.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 5.6 [3.0 to 9.7]

35. Secondary Outcome: Time to New Metastases: Phase I and Phase II
Description: Time to new metastasis was defined as the time from the ontorpacept infusion (Day 1 of Cycle 1) to a new lesion appearance. Participants without new lesion or participants with new metastases after 2 or more missing/inadequate disease assessment or participants with new metastases after the start date of alternate anti-cancer therapy were censored at their last response assessment date or last assessment prior to the start date of alternate anti-cancer therapy whichever was earlier.
Time Frame: Time from the first ontorpacept infusion (Day 1 of Cycle 1) until the appearance of new lesion or death or censoring date, whichever occurred first (maximum exposure up to 74.1 weeks for Phase I and 88 weeks for Phase II)
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Months | NA [7.9 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and full range of 95% CI could not be calculated as no participant had event. | NA [NA to NA] — Median and full range of 95% CI could not be calculated as no participant had event. | NA [6.0 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 4.7 [1.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [3.9 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events.

36. Secondary Outcome: Number of Participants With a Worsening of Eastern Cooperative Oncology Group (ECOG) Performance Status: Phase I and Phase II
Description: ECOG performance were classified as 5 grades: 0: fully active, able to carry on all pre-disease performance without restriction; 1: restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2: ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours; 3: capable of only limited selfcare, confined to bed or chair more than 50% of waking hours and 4: completely disabled, cannot carry on selfcare and totally confined to bed or chair. Higher score indicated lower health status. Worsening of ECOG was defined as a worsening from baseline (i.e., increase) in the ECOG assessment level and was recorded in two consecutive assessments.
Time Frame: From Baseline up to 30 Days post last dose of study treatment/start of new anti-cancer therapy whichever occurred first (maximum exposure upto 74.1 and 88 weeks; maximum follow up to approx. 78.1 and 92 weeks for Phase I and II respectively)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Participants | 0 | 0 | 0 | 6 | 2 | 4

37. Secondary Outcome: Number of Participants With a Worsening of Global Health Status / Quality of Life (QoL) Status: Phase I and Phase II
Description: QOL was assessed with European organisation for research and treatment of cancer (EORTC) QoL Questionnaire Core 30 (QLQ-C30) tool. The EORTC QLQ-C30 is self-administered, self-reported general cancer-specific questionnaire consisting of 30 items covered by one of 3 dimensions: global health status (2 items): functional scales(15 total items addressing either physical, emotional, cognitive/social functioning) and symptom scales(13 total items addressing either fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea/financial impact). Higher score indicated better overall QoL. Worsening of Global Health Status /QoL assessments was defined as at least a 10-point decrease from baseline in the standardized score (linear transformation) of Global Health Status/QoL.
Time Frame: as for outcome 36
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
Number analyzed (Participants) | 3 | 3 | 3 | 32 | 13 | 22
Participants | 2 | 2 | 2 | 17 | 9 | 12

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1up to 30 Days post last dose of study treatment or start of new anti-cancer therapy whichever occurs soonest (maximum exposure up to 74.1 and 88 weeks; maximum follow up to approx. 78.1 and 92 weeks for Phase I and II respectively)
Description: Same event may appear as both AE and SAE, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in another participant, or a participant may have experienced both SAE and non-SAE. SAS included all participants who were enrolled, allocated to treatment, and received at least one non-zero dose of study treatment.
Arm/Group | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B)
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 1/3 | 12/32 | 2/13 | 9/22
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 9/32 | 8/13 | 15/22
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 24/32 | 12/13 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin (N=3) | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin (N=3) | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin (N=3) | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) (N=32) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) (N=13) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiotoxicity (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Ontorpacept 0.2 mg/kg + Doxorubicin (N=3) | Phase I: Ontorpacept 0.7 mg/kg + Doxorubicin (N=3) | Phase I: Ontorpacept 2.0 mg/kg + Doxorubicin (N=3) | Phase II: Ontorpacept 0.2 mg/kg + Doxorubicin (Cohort A) (N=32) | Phase II: Ontorpacept 1.0 mg/kg + Doxorubicin (Cohort C) (N=13) | Phase II: Ontorpacept 2.0 mg/kg + Doxorubicin (Cohort B) (N=22)
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 20 | 9 | 14
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 12 | 5 | 6
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 11 | 6 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 7 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 2 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 5 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 4 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 1 | 22 | 9 | 15
Pyrexia (General disorders) | 0 | 0 | 2 | 5 | 2 | 2
Chills (General disorders) | 1 | 0 | 0 | 4 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 2 | 4
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 14 | 8 | 16
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 8 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 2 | 3
Platelet count decreased (Investigations) | 0 | 0 | 1 | 11 | 9 | 19
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 12 | 7 | 15
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 9 | 7 | 10
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 6 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 4 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 1 | 2 | 13 | 5 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 7 | 2 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 4 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 10 | 9 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 11 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 6 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 13 | 2 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 9 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 7 | 2 | 4
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 8 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 4 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 2 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 2 | 3
Vision blurred (Eye disorders) | 0 | 1 | 0 | 2 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04996004/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT04996004/SAP_001.pdf